CLINICAL TRIAL: NCT03314194
Title: Plant Based Diet, Ethnicity, and the Gut Microbiome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Seth Bordenstein (Unknown)
Responsible Party: Principal Investigator, Heidi J. Silver, Research Associate Professor of Medicine, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 171170
Record Dates: First submitted 2017-08-28; First posted 2017-10-19 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Diet Modification; Microbial Colonization
MeSH Terms: conditions — Communicable Diseases | interventions — Diet, Plant-Based

STUDY DESIGN:
Intervention Model Description: Pre Post Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Plant Based Diet Group (Experimental): Study aims for two cohorts of 20 females each, being tested over 6 days in two conditions: habitual diet versus plant based diet.
  Interventions: Other: Plant Based Diet

INTERVENTIONS:
Other: Plant Based Diet — Plant Based Diet for 4 Days Compared to Habitual Diet

SUMMARY:
Samples will be collected to determine human genetic variation, fecal and oral microbial communities, and metabolome products. Several evolutionary and ecological diversity metrics will be distilled to test: a) if microbiome variation within each ethnicity is less than that between ethnicities; b) if microbiome variation is finely structured according to genetic relatedness; and c) if dietary variation impacts human genome x microbiome associations.

DETAILED DESCRIPTION:
To characterize the human gut microbiome under highly controlled dietary intake in healthy normal weight adult participants who differ by ethnicity: White non-Hispanic and Black non-Hispanic adults. Samples will be collected to determine human genetic variation, fecal and oral microbial communities, and metabolome products. Several evolutionary and ecological diversity metrics will be distilled to test: a) if microbiome variation within each ethnicity is less than that between ethnicities; b) if microbiome variation is finely structured according to genetic relatedness; and c) if dietary variation impacts human genome x microbiome associations.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 18-40
* BMI 18.5-24.9
* Caucasian or African American

Exclusion Criteria:

* Not weight stable
* Using Medications
* Using Dietary Supplements
* Chronic Disease
* Tobacco Use
* Drug Use
* Pregnant or Lactating
* Diet Restrictions
* Vegetarian or Vegan

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Microbial Community Profile | 4 days
  A microbial community profile will be generated for each individual using high-throughput Illumina sequencing of the 16S rDNA microbial gene sequence. This community profile of each subjects microbiome will be assessed from a minimum of 10,000 sequences per individual at multiple timepoints. The profile will be used to quantify how inter-individual variation of the microbiome varies across ethnicities.

CONTACTS AND LOCATIONS:
Overall Officials: Heidi J Silver, Ph.D., Principal Investigator — Research Associate Professor
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
No Plan

REFERENCES:
- [Derived] Li J, George Markowitz RH, Brooks AW, Mallott EK, Leigh BA, Olszewski T, Zare H, Bagheri M, Smith HM, Friese KA, Habibi I, Lawrence WM, Rost CL, Ledeczi A, Eeds AM, Ferguson JF, Silver HJ, Bordenstein SR. Individuality and ethnicity eclipse a short-term dietary intervention in shaping microbiomes and viromes. PLoS Biol. 2022 Aug 23;20(8):e3001758. doi: 10.1371/journal.pbio.3001758. eCollection 2022 Aug. PMID 35998206